CLINICAL TRIAL: NCT07289828
Title: Prediction of Pre-existing Lower Extremity Injuries Using Lower Limb-worn Inertial Measurement Units
Brief Title: Prediction of Lower Extremity Injuries Using Lower Limb-worn Inertial Measurement Units
Acronym: PredKnee
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Christina Valle, Senior physician, Technical University of Munich
Other Study IDs: KneeInjuryPred
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lower Extremity Injuries
Keywords: prediction; ankle injury; knee injury; inertial sensor; artificial intelligence
MeSH Terms: conditions — Ankle Injuries; Knee Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- test group: All participants were sports students at TUM School of Medicine and Health. Of all participants, inertial sensor data were collected during walking and running on a defined track (5 minutes walking, 5 minutes running, 5 minutes walking on a standard 400 m oval tartan track). All participants completed questionnaires regarding previous injuries, comorbidities, sports activity, and preventive measures undertaken.
  Interventions: Other: IMU Data collection; Other: Questionnaire

INTERVENTIONS:
Other: IMU Data collection — Participants were walking and running while wearing inertial measurement units (IMU) on both legs. The IMUs (MetaMotionS sensor by Mbientlab) where recording at 100Hz (accelerometer and gyroscope) and 25Hz (magnetometer).
Other: Questionnaire — On the day of the examination, the test subjects completed a standardized questionnaire on previous injuries, type of sport, sporting activity, and preventive measures.

SUMMARY:
This study analyses questionnaires and inertial sensor data from 108 sports science students regarding previous lower extremity injuries, sports activity, and preventive measures, combined with the prospective development of an AI-based prediction algorithm.

Inertial sensor data were collected during walking and running on a standard 400 m track, with sensors placed on the thighs and ankles, and heart rate recorded via smartwatch. Participants also completed questionnaires on previous injuries, comorbidities, sports activity, and prevention.

The aim is to use the anonymized data to identify gait and running patterns associated with prior knee and ankle injuries using AI analysis, and to correlate these findings with sports activity and preventive measures.

Hypothesis: Prior lower extremity injuries leave specific gait and running patterns detectable by inertial sensors and AI-based analysis.

DETAILED DESCRIPTION:
In this study, analysis of questionnaires and inertial sensor data from 108 sports science students is conducted with regard to previous injuries of the lower extremities, their sports activities, and a possible association with performed preventive measures, along with the prospective development of an AI-based prediction algorithm to detect prior injuries of the lower extremities.

In all participants, inertial sensor data were collected during walking and running on a defined track (5 minutes walking, 5 minutes running, 5 minutes walking on a standard 400 m oval tartan track). Sensors were placed on the lateral aspects of both thighs above the knee joint and on the lateral aspects of both ankles above the lateral malleolus. In addition, participants wore a smartwatch on the left wrist to record heart rate. Furthermore, participants completed questionnaires regarding previous injuries, comorbidities, sports activity, and preventive measures undertaken.

The aim of the current analysis is to utilize the anonymized data from questionnaires and inertial sensors to identify gait and running patterns indicative of previous injuries of the lower extremities (knee and ankle) by means of an AI algorithm, and to correlate these findings with reported sports activities and preventive measures.

Hypothesis: Previous injuries of the lower extremities (particularly of the knee and ankle) result in specific gait and running patterns measurable by inertial sensors, which can be identified through AI-based analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjectively healthy participants
* Age: >18 years and under 60 years
* German language skills sufficient to follow the exercise instructions and complete the questionnaires

Exclusion Criteria:

* Age <18 years or >60 years
* Recent injuries and trauma to the lower extremities (less than 6 months ago)
* Acute malignant disease
* Acute inflammatory disease
* Lack of German language skills
* Lack of cardiopulmonary endurance for testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sport students at TUM School of Medicine and Health
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
IMU data | at baseline
  Time-stamped, unfiltered, device-coordinate-based 3-axis IMU data (Ax, Ay, Az) from four IMUs, placed laterally on both thighs (above the knee joint) and on both ankles (above the lateral malleolus).

SECONDARY OUTCOMES:
questionnaire injuries lower extremity | Baseline
  Participants reported previous injuries and illnesses affecting the lower extremities on a standardized questionnaire.
questionnaire sports activity | Baseline
  Participants indicated their sport and intensity level on a standardized questionnaire.
questionnaire prevention | baseline
  Participants indicated on a standardized questionnaire whether preventive measures to avoid sports injuries were being implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger von Eisenhart-Rothe, Prof. Dr. med., Study Director — Department of Orthopaedics and Sports Orthopaedics, TUM University Hospital
Locations (1):
- TUM University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
IDP is not permitted due to data protection regulations.